CLINICAL TRIAL: NCT01810978
Title: Efficacy of Synbiotics in Infants With Cyanotic Congenital Heart Disease
Brief Title: Synbiotics in Infants With Cyanotic Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Assoc Prof, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 128/01.10.2012
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease, probiotic, prebiotic
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Inulin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacterium lactis plus inulin (Active Comparator): Bifidobacterium lactis plus inulin
  Interventions: Dietary Supplement: Maltodextrin
- maltodextrin (Placebo Comparator): maltodextrin
  Interventions: Dietary Supplement: Bifidobacterium lactis plus inulin

INTERVENTIONS:
Dietary Supplement: Bifidobacterium lactis plus inulin — 5 billion unit Bifidobacterium lactis plus 900 mg inulin per day will be given
  Arms: maltodextrin
Dietary Supplement: Maltodextrin — same amount of maltodextrin per day will be given as placebo
  Arms: Bifidobacterium lactis plus inulin

SUMMARY:
Infants with congenital heart disease have more frequent infections and exposures to antibiotics than healthy infants. The investigators hypothesized that synbiotics may reduce the rate of sepsis and necrotizing enterocolitis in infants with CHD

DETAILED DESCRIPTION:
Infants with congenital heart disease have more frequent infections and exposures to antibiotics than healthy infants. Probiotics may prevent pathogen colonization in infants with CHD. Therefore, the investigators hypothesized that synbiotics may reduce the rate of sepsis and necrotizing enterocolitis in infants with CHD

ELIGIBILITY:
Inclusion Criteria:

* Cyanotic congenital heart disease
* infants >35 weeks of gestational age
* Born at or transferred to Sami Ulus CH

Exclusion Criteria:

* Congenital anomalies of the intestinal tract

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Sepsis | 8 weeks

SECONDARY OUTCOMES:
Necrotizing enterocolitis | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Banu Aydın, MD, Principal Investigator — MD
Locations (1):
- Sami Ulus CH, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Ellis CL, Rutledge JC, Underwood MA. Intestinal microbiota and blue baby syndrome: probiotic therapy for term neonates with cyanotic congenital heart disease. Gut Microbes. 2010 Nov-Dec;1(6):359-66. doi: 10.4161/gmic.1.6.14077. PMID 21468216
- [Derived] Dilli D, Aydin B, Zenciroglu A, Ozyazici E, Beken S, Okumus N. Treatment outcomes of infants with cyanotic congenital heart disease treated with synbiotics. Pediatrics. 2013 Oct;132(4):e932-8. doi: 10.1542/peds.2013-1262. Epub 2013 Sep 16. PMID 24043284
- See also: http://www.ncbi.nlm.nih.gov/pubmed/21468216 — http://www.ncbi.nlm.nih.gov/pubmed/21468216